CLINICAL TRIAL: NCT03716375
Title: A Randomized Controlled Study of Fibrinolytic Treatment for Purulent Pleural Effusion in Children
Brief Title: Efficacy of Fibrinolytic Agents in Complicated Pleural Effusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Baoping XU, Chief of Respiratory Department, Beijing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCHlung011
Record Dates: First submitted 2018-10-07; First posted 2018-10-23 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Complicated Pleural Effusion/ Empyema
Keywords: Pleural empyema, urokinase
MeSH Terms: conditions — Empyema, Pleural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- use of fibrinolytic agent (Experimental): Chest tube drainage with intrapleural urokinase instillation 1000 IU/ml
  Interventions: Drug: Intrapleural Medications
- no use of any drug (No Intervention): Chest tube drainage

INTERVENTIONS:
Drug: Intrapleural Medications — urokinase
  Arms: use of fibrinolytic agent

SUMMARY:
Intrapleural administration of fibrinolytic therapy, urokinase in parapneumonic effusion and empyema has been shown to decrease the need for surgical intervention and length of hospital stay. Pleural adhesions are easily formed in the early stages of empyema and the thickening of the pleural causes subsequent treatment difficulties. The goal of this study was to observe and compare the efficacy of treatment in empyema patients with urokinase and chest drainage or with chest drainage or with chest tube drainage alone so as to provide evidence for guiding clinical treatment.

DETAILED DESCRIPTION:
Empyema, a collection of pus in the pleural space has been continuously associated with morbidity and mortality rates of 10-20%. Increase in the incidence of empyema with change in pattern of disease and the causative organism has demonstrated a challenge in the diagnosis and treatment. In the recent years many studies and clinical trials have been done among adults and children regarding the optimal empyema treatment and its efficacy and some are still in the process of further study. Appropriate treatment according to the three stages of empyema (i.e. exudative stage, fibropurulent stage and organizing stage) has constantly been under frequent research, finding which treatment is more effective (i.e. antibiotics, chest tube drainage, intrapleural fibrinolytics, VATS and decortication alone in combination) and when is the proper time for intervention. Intrapleural instillation of urokinase was initially described in 1994 on pediatric population and since then lots of studies have been reported. Therefore, the investigators conducted a randomized controlled study with relevant inclusion and exclusion criteria to assess the success rate of intrapleural urokinase administration among the patients with Complicated Pleural Effusion (CPE) / empyema comparing it with drainage alone. All case patients in this study received antibiotic empirically or with sensitivity when microbiological tests available, chest tube drainage along with urokinase intrapleural therapy or drainage alone for treatment of CPE/empyema.

Patients will be randomized into two groups: one is chest tube drainage and intrapleural fibrinolytic agent and another is chest tube drainage alone. The group with intrapleural fibrinolytic agent will receive urokinase 10ml of 1000 IU/ml in children aged less than or equal to 1 year or 40ml of 1000 IU/ml in children aged more than 1 year and the other group with drainage alone. The first instillation of the agent is done at the time of chest tube insertion of 12Fr or 14Fr tube, after instillation the chest tube is closed for 4 hours. The chest tube is then unclamped after 4 hours and connected to the suction system with pressure of -20cm H2O for 8 hours and the process is repeated every 12 hourly. The procedure was done for 3 consecutive days and was evaluated with daily chest X-ray and followed chest tube removal when the drainage was less than 40ml/day or according to the clinical and radiological response of patients with treatment.

The trial is being done for 12 months with 80 participants taken from one center, Beijing children´s Hospital.

The aim of this study is to evaluate difference among intrapleural urokinase as the initial treatment for children with pleural empyema against chest tube drainage alone. Length of hospital stay, number of days chest tube drainage, number of days of fever after tube insertion, complications such bleeding, chest pain will be compared between the two groups.

ELIGIBILITY:
Pleural Empyema diagnostic criteria were based on the "Zhu Futang Practical Pediatrics" (the 7th Edition) and The American Thoracic Society consensus guidelines for management of empyema.

* Frank pus at tapping or organism demonstrated on Gram stain or culture
* Pleural fluid pH < 7.2, glucose < 60mg/dl, LDH>1000 IU/ml, protein > 3g/ml and white cells 15,000 cells/mm cube
* Physical, radiological and laboratory signs accompanying the relevant clinical picture

Inclusion Criteria:

* Previously healthy child with age between 1 month to 18 years
* Admitted with diagnosis of Pleural empyema requiring chest tube insertion and fibrinolytics (as judged by the attending physician) with the following criteria:

I. Pneumonia with pleural empyema based on chest ultrasound and CT scan. II. Need for further intervention based on clinical criteria (persistent fever despite antibiotics for at least 48 hours, significant respiratory distress, tachypnea or hypoxia as a result of pleural empyema.

Exclusion Criteria:

Subject will be excluded if she or he has one of the followings:

* Empyema as result of tuberculosis, fungus or noninfectious causes (e.g. malignancy)
* Known coagulation impairment
* Suspected allergy to urokinase
* Child has already undergone drainage procedure or drug was used in 30 days (e.g.

chest tube or VATS

* Chronic lung diseases or other chronic illnesses (e.g. Immunodeficiency, neurological impairment possible)
* Significant thoracic trauma in last 2 months
* Severe arterial hypertension
* Presence of Pneumothorax before treatment (i.e. bronchopleural fistula)
* Pregnancy
* Breast feeding
* Poor compliance
* Contraindication in the presence of fibrinolytic agent

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | 2 weeks

SECONDARY OUTCOMES:
Days of fever after chest tube insertion | 3 to 4 days
Duration of drainage | 2 weeks
Complications | 2weeks
  number of participants changed to open thoracotomy
Failure rate | 2weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xu Baoping, MD, PhD, Principal Investigator — Beijings Children´s Hospital of Capital Medical University, China

REFERENCES:
- [Result] Shirota C, Uchida H. Initial treatment of septated parapneumonic empyema with drainage plus fibrinolytic agents is equally effective as video-assisted thoracoscopic surgery, and is suitable as first-line therapy. Transl Pediatr. 2015 Jan;4(1):41-4. doi: 10.3978/j.issn.2224-4336.2015.02.01. PMID 26835359
- [Result] Stefanutti G, Ghirardo V, Barbato A, Gamba P. Evaluation of a pediatric protocol of intrapleural urokinase for pleural empyema: a prospective study. Surgery. 2010 Sep;148(3):589-94. doi: 10.1016/j.surg.2010.01.010. Epub 2010 Mar 20. PMID 20304453
- [Result] Walker W, Wheeler R, Legg J. Update on the causes, investigation and management of empyema in childhood. Arch Dis Child. 2011 May;96(5):482-8. doi: 10.1136/adc.2009.165357. Epub 2010 Aug 24. PMID 20736395